CLINICAL TRIAL: NCT01995500
Title: BioNIR Ridaforolimus Eluting Coronary Stent System (BioNIR) EUropean Angiography Study
Brief Title: Angiography Study of BioNIR Drug Eluting Stent System (NIREUS)
Acronym: NIREUS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medinol Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BioNIR-002
Record Dates: First submitted 2013-11-14; First posted 2013-11-26 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2020-05

CONDITIONS: Coronary Artery Stenosis
Keywords: CAD; PCI; ACS; non ACS; BioNIR; DES
MeSH Terms: conditions — Coronary Stenosis

STUDY DESIGN:
Intervention Model Description: This is a Drug-Device combination Product
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BioNIR (Experimental): The BioNIR Ridaforolimus Eluting Coronary Stent System is a single use device/drug combination product comprising:
  * Stent - a mounted Cobalt Chromium (CoCr) alloy based stent
  * Delivery System - Rapid Exchange (RX) Coronary System
  * Polymer matrix coating - Poly n-butyl methacrylate (PBMA) and CarboSil®
  * Ridaforolimus drug - CAS Registry Number: 572924-54-0 The drug Ridaforolimus is utilized on the stent system at a dose of 1.1 μg/mm2 (with a drug load of 100 μg per 2.75/3.00 x 17 mm stent).
  Interventions: Device: BioNIR
- Resolute (Active Comparator): The Endeavor Resolute Zotarolimus-Eluting Coronary Stent System consists of four subsystems:
  * Endeavor Resolute Stent - a premounted cobalt alloy based stent
  * Delivery system - Rapid Exchange (RX) Coronary System
  * Polymer system
  * Zotarolimus - drug The Resolute has a nominal drug dose of 1.6 µg zotarolimus per mm2 of the stent surface area.
  Interventions: Device: Resolute

INTERVENTIONS:
Device: BioNIR — drug-eluting stent
  Arms: BioNIR
Device: Resolute — drug-eluting stent
  Arms: Resolute

SUMMARY:
The NIREUS study aims to demonstrate angiographic non-inferiority for the BioNIR Ridaforolimus Eluting Coronary Stent System (hereafter referred to as BioNIR) in comparison to the Resolute zotarolimus-eluting stent (hereafter referred to as Resolute).

The trial hypothesis is that the BioNIR is non-inferior to the Resolute for the primary endpoint of angiographic in-stent late loss at 6 months.

DETAILED DESCRIPTION:
This is a prospective, multi-center, single-blind, two-arm, 2:1 randomized clinical trial.

Randomization will be stratified by the presence of medically treated diabetes vs. no medically treated diabetes and by site. Lesions planned to be treated must be declared and recorded at time of randomization.

Angiographic follow-up will be performed at 6 months. Clinical follow-up will be performed at 30 days, 6 months, and 1, 2, 3, 4, and 5 years post randomization.

The Primary Endpoint is in-stent late loss at 6 months as measured by the angiographic core laboratory.

Angiographic Secondary Endpoints to be evaluated at 6 months are:

* In-segment late loss
* Follow-up percent diameter stenosis (in-stent and in-segment)
* Binary restenosis (in-stent and in-segment)
* Length and patterns of angiographic restenosis (Mehran classification)

Clinical Secondary Endpoints to be evaluated at 30 days, 6 months, and 1, 2, 3, 4 and 5 years, except as noted, are:

* Device, Lesion, and Procedure Success at time of baseline procedure
* Target lesion failure (TLF; the composite of cardiac death, target vessel-related MI, or ischemia-driven TLR)
* Major adverse cardiac events (MACE; the composite rate of cardiac death, any MI or ischemia-driven TLR)
* Target vessel failure (TVF; the composite rate of death, target vessel-related MI, or ischemia-driven TVR)
* Overall Mortality
* Cardiac Death
* Myocardial Infarction
* Target Vessel Related MI
* Ischemia-driven TLR
* Ischemia-driven TVR
* Stent Thrombosis (ARC definite and probable)

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patient with an indication for PCI including angina (stable or unstable), silent ischemia (in absence of symptoms a visually estimated target lesion diameter stenosis of ≥70%, a positive non-invasive stress test, or FFR ≤0.80 must be present), NSTEMI, or recent STEMI. For STEMI the time of presentation to the first treating hospital, whether a transfer facility or the study hospital, must be >24 hours prior to randomization and enzyme levels (CK-MB or Troponin) demonstrating that either or both enzyme levels have peaked.
* Non-target vessel PCI are allowed prior to randomization depending on the time interval and conditions as follows:

  a. During Baseline Procedure: i. PCI of non-target vessels performed during the baseline procedure itself immediately prior to randomization if successful and uncomplicated defined as: <50% visually estimated residual diameter stenosis, TIMI Grade 3 flow, no dissection ≥ NHLBI type C, no perforation, no persistent ST segment changes, no prolonged chest pain, no TIMI major or BARC type 3 bleeding.

  b. Less than 24 hours prior to Baseline Procedure: i. Not allowed (see exclusion criteria #3). c. 24 hours-30 days prior to Baseline Procedure: i. PCI of non-target vessels 24 hours to 30 days prior to randomization if successful and uncomplicated as defined above.

ii. In addition, in cases where non-target lesion PCI has occurred 24-72 hours prior to the baseline procedure, at least 2 sets of cardiac biomarkers must be drawn at least 6 and 12 hours after the non-target vessel PCI. If cardiac biomarkers are initially elevated above the local laboratory upper limit of normal, serial measurements must demonstrate that the biomarkers are falling.

d. Over 30 days prior to Baseline Procedure: iii. PCI of non-target vessels performed greater than 30 days prior to procedure whether or not successful and uncomplicated.

* Patient or legal guardian is willing and able to provide informed written consent and comply with follow-up visits and testing schedule.

Angiographic inclusion criteria (visual estimate):

* Treatment of up to three de novo target lesions, maximum of one de novo target lesion per vessel
* Target lesion(s) must be located in a native coronary artery with visually estimated diameter of ≥2.5 mm to ≤4.25 mm and diameter stenosis ≥50% to <100%.
* Lesion must be ≤28 mm long and can be covered by a single study stent with maximum length of 33 mm (note: multiple focal stenoses may be considered as a single lesion and be enrolled if they can be completely covered with one stent).
* TIMI flow 2 or 3
* If more than one target lesion will be treated, the RVD and lesion length of each must meet the above criteria.

Exclusion Criteria:

* Planned procedures after the baseline procedure in either the target or non-target vessels.
* STEMI within 24 hours of initial time of presentation to the first treating hospital, whether at a transfer facility or the study hospital or in whom enzyme levels (either CK-MB or Troponin)have not peaked.
* PCI within the 24 hours preceding the baseline procedure and randomization.
* Non-target lesion PCI in the target vessel within 12 months of the baseline procedure.
* History of stent thrombosis.
* Cardiogenic shock (defined as persistent hypotension (systolic blood pressure <90 mm/Hg for more than 30 minutes) or requiring pressors or hemodynamic support, including IABP.
* Known LVEF <30%.
* Subject is intubated.
* Relative or absolute contraindication to DAPT for 12 months (including planned surgeries that cannot be delayed, or subject is indicated for chronic oral anticoagulant treatment).
* Hemoglobin <10 g/dL.
* Platelet count <100,000 cells/mm3 or >700,000 cells/mm3.
* White blood cell (WBC) count <3,000 cells/mm3.
* Clinically significant liver disease.
* Renal disease as defined by an estimated creatinine clearance <40 mL/min using Cockcroft-Gault equation.
* Active peptic ulcer or active bleeding from any site.
* Bleeding from any site within the prior 8 weeks requiring active medical or surgical attention.
* History of bleeding diathesis or coagulopathy or likely to refuse blood transfusions.
* If femoral access is planned, significant peripheral arterial disease which precludes safe insertion of a 6F sheath.
* Cerebrovascular accident or transient ischemic attack within the past 6 months, or any permanent neurologic defect attributed to CVA.
* Known allergy to the study stent components, whether in the BioNIR or Resolute, e.g. cobalt, nickel, chromium, molybdenum, Carbosil®, PBMA, Biolinx polymer, or limus drugs (ridaforolimus, zotarolimus, tacrolimus, sirolimus, everolimus, or similar drugs or any other analogue or derivative or similar compounds).
* Known allergy to protocol-required concomitant medications such as aspirin, or DAPT (clopidogrel, prasugrel, ticagrelor), or heparin and bivalirudin, or iodinated contrast that cannot be adequately pre-medicated.
* Any co-morbid condition that may cause non-compliance with the protocol (e.g. dementia, substance abuse, etc.) or reduced life expectancy to <24 months (e.g. cancer, severe heart failure, severe lung disease).
* Patient is participating in or plans to participate in any other investigational drug or device clinical trial that has not reached its primary endpoint.
* Women who are pregnant or breastfeeding (women of child-bearing potential must have a negative pregnancy test within one week before treatment).
* Women who intend to become pregnant within 12 months after the baseline procedure (women of child-bearing potential who are sexually active must agree to use a reliable method of contraception from the time of screening through 12 months after the baseline procedure).
* Patient has received an organ transplant or is on a waiting list for an organ transplant.
* Patient is receiving or scheduled to receive chemotherapy within 30 days before or any time after the baseline procedure.
* Patient is receiving oral or intravenous immunosuppressive therapy or has known life-limiting immunosuppressive or autoimmune disease (e.g., HIV). Corticosteroids are allowed.

Angiographic Exclusion Criteria (visual estimate):

* Unprotected left main lesions ≥30%, or planned left main intervention.
* Stenting of ostial LAD or LCX lesions (stenting of any diseased segment within 5 mm of the unprotected left main coronary artery).
* Lesions located within an arterial or saphenous vein graft or distal to a diseased arterial or saphenous vein graft.
* Moderately or heavily calcified lesions.
* Moderately or heavily tortuous or angulated lesions or vessels.
* Bifurcation lesions in the presence of a side branch ≥2.0 mm in diameter.
* Lesions containing thrombus.
* Total occlusions.
* In-stent restenotic lesions or lesions present within 10 mm of a previously implanted stent.
* Lesions requiring pre-dilatation with any device other than simple balloon angioplasty (e.g. atherectomy or cutting/scoring balloons).
* Another lesion in the target vessel is present that requires or has a high probability of requiring PCI during the baseline procedure or within 6 months after the baseline procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2014-03-19 (Actual); Primary Completion 2015-03-19 (Actual); Study Completion 2020-06-17 (Actual)

PRIMARY OUTCOMES:
In-stent late loss | 6 months
  In-stent late loss as measured by the angiographic core laboratory

SECONDARY OUTCOMES:
In-segment late loss | 6 months
  angiographic secondary endpoint
Follow-up percent diameter stenosis | 6 months
  angiographic: Follow-up percent diameter stenosis (in-stent and in-segment)
Binary restenosis | 6 months
  angiographic: Binary restenosis (in-stent and in-segment)
Length and patterns of angiographic restenosis | 6 months
  angiographic: Mehran classification
Device, Lesion, and Procedure Success | Determined at time of baseline procedure
  Device success is defined as achievement of a final in-stent residual diameter stenosis of <50% (by QCA), using the assigned device only and without a device malfunction.
  Lesion success is defined as achievement of a final in-stent residual diameter stenosis of <50% (by QCA) using any percutaneous method.
  Procedure success is defined as achievement of a final in-stent diameter stenosis of <50% (by QCA) using the assigned device and/or with any adjunctive devices, without the occurrence of cardiac death, Q wave or non-Q wave MI, or repeat revascularization of the target lesion during the hospital stay.
Target lesion failure | 30 days, 6 months, and 1, 2, 3, 4 and 5 years
  Clinical: TLF, the composite of cardiac death, target vessel-related MI, or ischemia-driven TLR
Major Adverse Cardiac Events (MACE) | 30 days, 6 months, and 1, 2, 3, 4 and 5 years
  Clinical: MACE, the composite rate of cardiac death, any MI or ischemia-driven TLR
Target vessel failure | 30 days, 6 months, and 1, 2, 3, 4 and 5 years
  TVF, the composite rate of death, target vessel-related MI, or ischemia-driven TVR
Overall Mortality | 30 days, 6 months, and 1, 2, 3, 4 and 5 years
  Clinical: Overall mortality during the trial period
Cardiac death | 30 days, 6 months, and 1, 2, 3, 4 and 5 years
  Clinical measure: The number of patients who suffered cardiac death
Myocardial Infarction | 30 days, 6 months, and 1, 2, 3, 4 and 5 years
  Clinical: myocardial infarction
Target vessel related MI | 30 days, 6 months, and 1, 2, 3, 4 and 5 years
  clinical: target vessel related MI
Ischemia driven TLR and TVR | 30 days, 6 months, and 1, 2, 3, 4 and 5 years
  clinical: TLR and TVR
Stent Thrombosis | 30 days, 6 months, and 1, 2, 3, 4 and 5 years
  clinical: Stent Thrombosis (ARC definite and probable)

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Hebrew University Medical Center, Jerusalem, Israel

REFERENCES:
- [Derived] Paradies V, Ben-Yehuda O, Jonas M, Banai S, Iniguez A, Perlman GY, Kandzari DE, Stone GW, Smits PC. A prospective randomised trial comparing the novel ridaforolimus-eluting BioNIR stent to the zotarolimus-eluting Resolute stent: six-month angiographic and one-year clinical results of the NIREUS trial. EuroIntervention. 2018 May 20;14(1):86-93. doi: 10.4244/EIJ-D-17-00890. PMID 29537374